CLINICAL TRIAL: NCT02919696
Title: A Phase 1 Study of Abemaciclib in Native Chinese Patients With Advanced and/or Metastatic Cancers
Brief Title: A Study of Abemaciclib (LY2835219) in Native Chinese Participants With Advanced and/or Metastatic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15531; I3Y-CR-JPBR (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2019-12-01

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: CDK4/6 Inhibitor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abemaciclib Dose Level 1 (Experimental): Abemaciclib 150 milligram (mg) administered every 12 hours, orally, cycle 1 and then in cycle 2. Participants may continue to receive treatment until discontinuation criteria are met. One cycle is defined as 28 days. (Cycle 1: 32 days), with modifications during Cycle 1 to enable pharmacokinetic (PK) sampling following a single dose and repeated doses.
  Interventions: Drug: Abemaciclib
- Abemaciclib Dose Level 2 (Experimental): Abemaciclib 200 mg administered every 12 hours, orally, cycle 1 and then in cycle 2. Participants may continue to receive treatment until discontinuation criteria are met. One cycle is defined as 28 days. (Cycle 1: 32 days), with modifications during Cycle 1 to enable PK sampling following a single dose and repeated doses.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219

SUMMARY:
The purpose of this study is to determine the safety of the study drug known as abemaciclib in native Chinese participants with advanced and/or metastatic cancers.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have histological or cytological evidence of cancer which is advanced and/or metastatic, and is an appropriate candidate for experimental therapy in the judgment of the investigator, after available standard therapies have ceased to provide clinical benefit.
* Have the presence of measureable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Are native Chinese men or women.
* Have adequate organ function, including:

  * Hematologic: Absolute neutrophil count (ANC) ≥1.5 x 109/Liters (L), platelets ≥100 x 109/L, and hemoglobin ≥9 grams per deciliter. Participants may receive erythrocyte transfusions to achieve this hemoglobin level or platelet transfusions to achieve platelet levels at the discretion of the investigator; however, initial study drug treatment must not begin earlier than the day after transfusion.
  * Hepatic: Bilirubin ≤1.5 times upper limits of normal (ULN), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤3.0 times ULN.
  * Renal: Serum creatinine ≤1.2 milligrams per deciliter (mg/dL) for males or ≤1.0 mg/dL for females.
* Have a performance status ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Recovered from the acute effects of therapy (treatment- related toxicity resolved to baseline) except for residual alopecia.
* Have an estimated life expectancy of ≥12 weeks.

Exclusion Criteria:

* Have received previous therapies for cancer (including chemotherapy, radiotherapy, immunotherapy, and investigational therapy) within 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug.
* Have an acute leukemia or other relevant cancers at the discretion of the investigator.
* Females who are pregnant or lactating.
* Participants consuming drugs or foods that are known to be inducers (for example, grapefruit juice, phenytoin, carbamazepine) or strong inhibitors of CYP3A4 should be excluded during Cycle 1.
* Have history or evidence of central nervous system (CNS) malignancy or metastasis. Screening of asymptomatic participants without history of CNS metastases is not required for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- China (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Yang N, Ji D, Shen W, Li W, Han R, Wang N, Tao H, Chapman SC, Sykes AK, Zhang W, Hu X. A Randomized Phase I Study of Abemaciclib in Chinese Patients with Advanced and/or Metastatic Cancers. Target Oncol. 2021 Mar;16(2):177-187. doi: 10.1007/s11523-020-00789-9. Epub 2021 Jan 25. PMID 33492568

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed were those who had progressive disease or died due to any cause while on treatment. Pharmacokinetic (PK) samples were collected at lower doses during cycle 1.
Groups:
- Abemaciclib 150 mg: Abemaciclib 150 milligram (mg) administered every 12 hours, orally, cycle 1 and then in cycle 2. Participants may continue to receive treatment until discontinuation criteria are met.
  One cycle is defined as 28 days. (Cycle 1: 32 days), with modifications during Cycle 1 to enable PK sampling following a single dose and repeated doses.
- Abemaciclib 200 mg: Abemaciclib 200 mg administered every 12 hours, orally, cycle 1 and then in cycle 2. Participants may continue to receive treatment until discontinuation criteria are met.
  One cycle is defined as 28 days. (Cycle 1: 32 days), with modifications during Cycle 1 to enable PK sampling following a single dose and repeated doses.
Period: Overall Study
Arm/Group | Abemaciclib 150 mg | Abemaciclib 200 mg
Started | 12 | 14
Received at Least One Dose of Study Drug | 12 | 13
PK 100 mg Abemaciclib Dose | 5 | 0
PK 150 mg Abemaciclib Dose | 0 | 2
Death On Treatment | 1 | 0
Progressive Disease | 7 | 9
Completed | 8 | 9
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Sponsor Decision | 1 | 1
Not completed — Never Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abemaciclib 150 mg | Abemaciclib 200 mg | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.58 (11.47) | 52.00 (8.76) | 53.72 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 13 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug Related Adverse Events
Description: Number of participants with one or more drug related adverse events. Clinically significant events were defined as serious adverse events, regardless of causality. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through End of Study (Up to 10 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 12 | 13
Participants | 12 | 13

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Abemaciclib and Its Metabolites Single Dose
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Abemaciclib and its Metabolites following a single oral dose.
Time Frame: Cycle 1, Day(D)1; Predose, 1, 4, 6, 8, 10, 24, 48 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 12 | 13
nanogram/milliliter (ng/mL) | 204 (70) | 210 (65)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of Abemaciclib and Its Metabolites (Twice Daily Dosing)
Description: PK: Maximum Concentration (Cmax) of Abemaciclib and its Metabolites following a twice daily dosing.
Time Frame: Cycle 1, Day(D) 31; Predose, 1, 2, 4, 6, 8, 10, 24 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Abemaciclib 100 mg: Abemaciclib 100 mg administered every 12 hours, orally, during cycle 1. Participants may continue to receive treatment until discontinuation criteria are met. One cycle is defined as 28 days. (Cycle 1: 32 days), with modifications during Cycle 1 to enable PK sampling following a single dose and repeated doses.
Arm/Group | Abemaciclib 100 mg | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 4 | 7 | 10
ng/mL | 205 (64) | 267 (71) | 320 (91)

4. Secondary Outcome: PK: Area Under Concentration Time Curve (AUC) From Time Zero to 12 Hours (AUC [0-12]) of Abemaciclib and Its Metabolites Single Dose
Description: PK: Area Under Concentration Time Curve (AUC) from Time Zero to 12 hours (AUC [0-12]) of Abemaciclib and its Metabolites following a single oral dose.
Time Frame: Cycle 1, Day(D)1; Predose, 1, 4, 6, 8, 10, 24, 48 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- Abemaciclib 150 mg: Abemaciclib 150 mg administered every 12 hours, orally, cycle 1 and then in cycle 2. One cycle is defined as 28 days. (Cycle 1: 32 days), with modifications during Cycle 1 to enable PK sampling following a single dose and repeated doses.
Arm/Group | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 12 | 13
nanogram*hour/milliliter (ng*hr/mL) | 1700 (75) | 1740 (68)

5. Secondary Outcome: PK: AUC From Time Zero to 12 Hours (AUC [0-12]) of Abemaciclib and Its Metabolites (Twice Daily Dosing)
Description: PK: AUC from Time Zero to 12 hours (AUC [0-12]) of Abemaciclib and its Metabolites following twice daily dosing
Time Frame: Cycle 1, Day(D) 31; Predose, 1, 2, 4, 6, 8, 10, 24 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Abemaciclib 100 mg | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 4 | 7 | 10
ng*hr/mL | 2190 (65) | 2770 (73) | 3270 (101)

6. Secondary Outcome: PK: AUC From Time Zero to Infinity (AUC[0-inf]) of Abemaciclib and Its Metabolites Single Dose
Description: PK: AUC from Time Zero to Infinity (AUC[0-inf]) of Abemaciclib and its Metabolites following a single oral dose.
Time Frame: Cycle 1, Day(D)1; Predose, 1, 4, 6, 8, 10, 24, 48 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 12 | 13
ng*hr/mL | 6790 (63) | 7580 (74)

7. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With a Complete Response (CR) or Partial Response (PR)
Description: ORR was defined as the percentage of randomized participants with a best overall response of complete response (CR) or partial response (PR) using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. Participants with unevaluable or unknown response status are considered nonresponders. Complete response (CR) is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. Partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions and no appearance of new lesions. Progressive disease (PD) is defined as at least a 20% increase in the sum LD of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) and the 20% increase must be at least one lesion must increase by an absolute value of ≥5 mm to be considered progression.
Time Frame: Baseline to Measured Progressive Disease (Up to 13 Months )
Population: All randomized participants who received at least one dose of study drug and had PR/CR data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 12 | 13
percentage of participants | 8.3 [0.2 to 38.5] | 7.7 [0.2 to 36.0]

ADVERSE EVENTS:
Time Frame: Up to 10 Months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Abemaciclib 150 mg | Abemaciclib 200 mg
All-Cause Mortality (participants affected / at risk) | 6/12 | 1/13
Serious Adverse Events (participants affected / at risk) | 2/12 | 4/13
Other Adverse Events (participants affected / at risk) | 12/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib 150 mg (N=12) | Abemaciclib 200 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib 150 mg (N=12) | Abemaciclib 200 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 5 (7)
Leukopenia (Blood and lymphatic system disorders) | 2 (7) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (6) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (24) | 11 (32)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (10)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (8) | 4 (9)
Influenza like illness (General disorders) | 2 (2) | 4 (6)
Localised oedema (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 7 (10) | 6 (8)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 4 (4)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (6) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 1 (1)
Bilirubin conjugated increased (Investigations) | 4 (4) | 1 (1)
Blood bilirubin increased (Investigations) | 4 (4) | 1 (1)
Blood bilirubin unconjugated increased (Investigations) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 6 (7) | 8 (11)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (23) | 8 (20)
Occult blood (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 4 (5) | 5 (6)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1)
White blood cell count decreased (Investigations) | 8 (17) | 6 (12)
Decreased appetite (Metabolism and nutrition disorders) | 10 (11) | 6 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT02919696/SAP_000.pdf
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT02919696/Prot_001.pdf